CLINICAL TRIAL: NCT06151028
Title: An Observational Study of Menopausal Symptom in Patients With Gynecological Malignancy After Oophorectomy (Carnation1)
Brief Title: An Observational Study of Menopausal Symptom in Patients With Gynecological Malignancy After Oophorectomy
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Ying Zhou
Record Dates: First submitted 2023-11-03; First posted 2023-11-30 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-10

CONDITIONS: Gynecological Malignancies; Menopausal Symptoms; Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual Blood, Urine, Fecal, Saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an observational study and did not involve interventions.

SUMMARY:
Through long-term dynamic monitoring of gynecologic malignant tumor patients undergoing early menopause after ovaries resection in our center, we explored the changes in menopausal symptoms and bone health status of this population, and studied the effects of platinum combined chemotherapy drugs on menopausal symptoms and bone loss in gynecologic malignant tumor patients. To find the optimal time point and effective regimen for MHT in gynecologic malignancies undergoing surgical menopause, and to provide guidance for osteoporosis screening and prevention strategies in women with gynecologic cancer.

DETAILED DESCRIPTION:
Gynecological malignancies are affecting the health of more and more women in the world, and the age of onset is also gradually younger. For women of reproductive age with gynecologic malignancies, surgery involving bilateral ovariectomy, followed by chemoradiotherapy or anti-estrogen therapy to maintain endocrine therapy, can lead to early menopause, leading to earlier and more severe menopausal syndrome and bone loss. Unlike the management of healthy women with natural menopause, the management of prognosis and quality of life in cancer patients with early menopause resulting from surgery combined with adjuvant therapy is more challenging and specific, and it is critical to identify management options for this complex patient population.

This study aims to conduct long-term dynamic monitoring of patients with gynecologic malignancies undergoing early menopause after ovaries resection in our center, explore the changes in menopausal symptoms and bone health status of this population, and study the effects of platinum combined chemotherapy drugs on menopausal symptoms and bone loss in patients with gynecologic malignancies. To find out the best time point and effective program of menopausal hormone therapy for gynecological malignant tumor patients with surgical menopause, and provide guidance for osteoporosis screening and prevention strategies for women with gynecological cancer.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with gynecological malignancies aged 18-55 years old;

  * Tumor types include endometrial cancer, cervical cancer, epithelial ovarian cancer;

    * All patients received standard stage operation and treatment;

      * Patients with bilateral ovaries resection; ⑤Voluntarily participate in this study, willing to sign informed consent, and have long-term follow-up conditions.

Exclusion Criteria:

* Menopause (women over 40 years of age stop menstruation for 12 months, excluding pregnancy and other diseases that may cause amenorrhea can be clinically diagnosed as menopause); Or AMH < 0.2ng/ml (China Menopause Management and Menopause Hormone Therapy Guidelines 2023 edition); Or FSH> 40 mIU/ml after two checks within one month;

  * Other tumors were combined within 2 years and were still in radiotherapy, chemotherapy or hormone therapy;

    * Diagnosis of immunodeficiency disease or active hepatitis B, C, active tuberculosis; ④Serious organic diseases of the organs, etc., can not cooperate with the study follow-up; ⑤Long-term use of hormonal drugs for rheumatic system diseases, such as glucocorticoids;

      * Patients who have previously received pelvic or abdominal radiotherapy; ⑦ ECOG score ≥3 points; ⑧The patient did not sign informed consent or was unwilling to accept follow-up interviews.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study is an observational study. It is expected that the department will receive about 3000 patients with gynecologic malignancies in the next 10 years. Based on this, we plan to collect 490 premenopausal patients with gynecologic malignancies from the First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital) during 2023.12~2033.12. All enrolled patients underwent standard tumor staging or tumor cell reduction involving bilateral ovariectomy and completed follow-up therapy (observation or chemotherapy) according to NCCN guidelines. The enrolled patients were followed up regularly for tumor risk assessment, menopause scale assessment, bone health assessment and related imaging examination. The medical history and data were complete.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Bone mineral density was followed up at 1, 2, 3, 6, 9, 12, 24 and 36 months after the operation
  Bone density examination
KMI | The scale was evaluated at 1, 3, 6 and 12 months after surgery.
  Modified Kupperman Index（0-63score）
MENQOL | The scale was evaluated at 1, 3, 6 and 12 months after surgery.
  Menopause-Specific Quality of Life（0-174score）
HADS | The scale was evaluated at 1, 3, 6 and 12 months after surgery.
  Hospital Anxiety and Depression Scale（0-21score）
IOF | The scale was evaluated at 1, 3, 6 and 12 months after surgery.
  Osteoporosis Risk one-minute Test Scale (Yes or No)
PSQI | The scale was evaluated at 1, 3, 6 and 12 months after surgery.
  Pittsburgh sleep quality index（0-21score）

SECONDARY OUTCOMES:
OS | 5 year
  OS was defined as the time interval between a patient's diagnosis of gynecologic malignancy and death from any cause or the end of the last follow-up date.
PFS | 5 year
  PFS is defined as the time interval between a patient's diagnosis of gynecological malignancy and the first occurrence of progression of the disease or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhou, MD, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No